CLINICAL TRIAL: NCT06040346
Title: A Phase 2a, Multicenter, Open-label, Dose-finding, Dose Escalation Study of Meplazumab in Adult Patients Diagnosed with Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Open-Label Study to Assess Meplazumab in Adult Patients Diagnosed with Plasmodium Falciparum
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Pacific Meinuoke Bio Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MPZ-MAL-01
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — meplazumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Groups (Experimental): Up to 60 participants will be enrolled into 1 of 3 meplazumab dose levels (20 participants/dose level).
  Interventions: Drug: Meplazumab for Injection

INTERVENTIONS:
Drug: Meplazumab for Injection — Meplazumab, an erythrocytic stage-macromolecular antibody drug, has the potential to control clinical occurrence of falciparum malaria. Meplazumab is a humanized anti-CD147 immunoglobulin G subclass 2 (IgG2) monoclonal antibody with strong affinity to CD147. CD147 is expressed on erythrocyte lineage cells throughout erythroid development, including mature erythrocytes and is the target for Plasmodium merozoites to allow reorientation and subsequent invasion of the erythrocytes.

SUMMARY:
This phase 2a open-label study to assess Meplazumab in adult patients diagnosed with Plasmodium falciparum

DETAILED DESCRIPTION:
Rationale:

Meplazumab, an erythrocytic stage-macromolecular antibody drug, has the potential to control clinical occurrence of falciparum malaria. Meplazumab is a humanized anti-CD147 immunoglobulin G subclass 2 (IgG2) monoclonal antibody with strong affinity to CD147. CD147 is expressed on erythrocyte lineage cells throughout erythroid development, including mature erythrocytes and is the target for Plasmodium merozoites to allow reorientation and subsequent invasion of the erythrocytes. Nonclinical studies have demonstrated that meplazumab binding to CD147 interferes with the receptor-ligand interaction between CD147 and rhoptry-associated protein 2 (RAP2) of the P. falciparum merozoite and inhibits the formation of parasitophorous vacuoles of P. falciparum thus preventing the invasion of P. falciparum into human erythrocytes. Furthermore, the therapeutic and prophylactic effects of meplazumab were demonstrated in vivo using a human erythrocyte chimeric NOG mouse model, which is considered as an optimal choice for in vivo inhibition efficacy study for human-hosted P. falciparum.

Meplazumab has previously been studied in healthy participants in two Phase 1 studies and has also been evaluated for activity in 2 completed clinical trials in patients diagnosed with coronavirus disease 2019 (COVID 19). In the safety, tolerability, and pharmacokinetics study in healthy participants, MPZ I-01, results demonstrated a high and prolonged receptor occupancy (RO%) of meplazumab at CD147.

This Phase 2a study is designed as a dose escalation trial to assess safety of meplazumab in the target population and to evaluate whether meplazumab is efficacious in treating malaria. The data obtained in this study will be used to determine a recommended meplazumab dose for future Phase 2b and 3 efficacy trials.

Overall Design:

This is a Phase 2a multicenter, open-label, dose-finding, dose escalation study. The study will recruit participants with confirmed P. falciparum infection. Up to 60 participants will be enrolled into 1 of 3 meplazumab dose levels (20 participants /dose level).

Number of Participants:

Up to 60 participants will be enrolled into 1 of 3 meplazumab dose levels (20 participants/dose level).

Intervention Groups and Duration:

Participants will be administered a single intravenous (IV) infusion dose of meplazumab 120±5 minutes on Day 0 and confined for 72 hours after dosing (up to Day 3) to monitor for safety and tolerability of therapy, and to ensure treatment response. During confinement, blood sampling for safety, pharmacokinetic (PK), and RO pharmacodynamic (PD) testing at predefined times will be collected as specified per the Schedule of Assessment (SoA). Furthermore, in a subset of 10 participants/dose level, additional (serial) PK and PD sample will be collected at 1, 2, 4 and 8 hours post end-of-infusion. Up to 3 additional samples may be added to the Day 0-3 serial sample collection period.

If clinically well, participants may be discharged from the clinical unit on Day 3 at the Investigator's discretion. Participants will return to the study center for follow-up visits on Days 28±2, 56±7, 84±7 and 182±7 (End of Study) for safety, tolerability, PK, PD (RO rate), and immunogenicity assessments as per the SoA (Weeks 4, 8, 12 and 26).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent signed by the study participant or legally authorized representative
2. Adults 18 to 55 years at the time of signing the informed consent form (ICF)
3. Female participants are eligible to participate if they do not qualify as a woman of childbearing potential (WOCBP), as defined in Section 10.4.
4. Male participants who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in Section 10.4.
5. BMI ≥18 to ≤30 kg/m2
6. Mono-infection with P. falciparum documented by:

   * Microscopically confirmed parasite infection using by Giemsa-stained thick film (refer to the laboratory manual for details) consisting of 1000 - 100,000 asexual parasites /µL of blood and
   * Documented fever (≥38.0°C oral, rectal or tympanic; ≥37.5°C axillary) or documented history of fever in previous 24 hours

Exclusion Criteria:

1. Presence of severe malaria (as defined by World Health Organization Guidelines for Malaria 16 February 2021).

   • Severe falciparum malaria is defined as one or more of the following, occurring in the absence of an identified alternative cause and in the presence of P. falciparum asexual parasitemia.
   * Impaired consciousness: A Glasgow coma score <11 in adults
   * Prostration: Generalized weakness so that the person is unable to sit, stand or walk without assistance
   * Multiple convulsions: More than 2 episodes within 24 h
   * Acidosis: A base deficit of >8 mEq/L or, if not available, a plasma bicarbonate level of <15 mmol/L or venous plasma lactate ≥5 mmol/L. Severe acidosis manifests clinically as respiratory distress (rapid, deep, labored breathing).
   * Hypoglycemia: Blood or plasma glucose <2.2 mmol/L (<40 mg/dL)
   * Severe malarial anemia: Hemoglobin concentration ≤7 g/dL or a hematocrit of ≤20% in adults with a parasite count >10,000/μL
   * Renal impairment: Plasma or serum creatinine >265 μmol/L (3 mg/dL) or blood urea >20 mmol/L
   * Jaundice: Plasma or serum bilirubin >50 μmol/L (3 mg/dL) with a parasite count >100,000/ μL
   * Pulmonary edema: Radiologically confirmed or oxygen saturation <92% on room air with a respiratory rate >30/min, often with chest indrawing and crepitations on auscultation
   * Significant bleeding: Including recurrent or prolonged bleeding from the nose, gums or venepuncture sites; hematemesis or melena
   * Shock: Compensated shock is defined as capillary refill ≥3 s or temperature gradient on leg (mid to proximal limb), but no hypotension. Decompensated shock is defined as systolic blood pressure <80 mmHg in adults, with evidence of impaired perfusion (cool peripheries or prolonged capillary refill).
   * Hyperparasitemia: P. falciparum parasitemia >10%
2. Antimalarial treatment (alone or in combination) during the following periods before Screening:

   * Piperaquine, mefloquine, naphthoquine or sulfadoxine-pyrimethamine within 6 weeks prior to Screening.
   * Amodiaquine, chloroquine within 4 weeks prior to Screening.
   * Any artemisinin derivative (artesunate, artemether or dihydroartemisinin), quinine, lumefantrine or any other antimalarial treatment or antibiotic with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones and azithromycin) within 14 days prior to Screening.
   * Any herbal products or traditional medicines, within the past 7 days.
3. Previous participation in any malaria vaccine study or received malaria vaccine within 3 months of Screening Visit.
4. Known allergy to any study medication, including allergy to any component of protocol prescribed rescue treatment i.e., country-specific ACT regimen.
5. Any clinically important illness, including but not limited to a history of clinically significant chronic respiratory disease (eg, chronic obstructive pulmonary disease [COPD] or asthma), medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product.
6. Participants participate in another clinical study. There will be a need for washout with 5 half-lives depending on the study treatment or 30 days, whichever is longer.
7. Use of anti-cancer, anti-transplant rejection, or immunomodulatory biological drug or kinase inhibitor (e.g., tocilizumab, sarilumab) or Janus kinase inhibitors (within 30 days of enrollment or 5 times the half-life [whichever is longer]).
8. Chronic corticosteroids use equivalent to daily oral prednisone >10 mg per day (10 mg oral prednisone every other day is allowed).
9. Live (live-attenuated) vaccines are not permitted within 2 weeks prior to study treatment or during the study treatment and safety follow-up periods.
10. Presence of Hepatitis A IgM, Hepatitis B surface antigen, or Hepatitis C antibody.
11. TBL >1.5 × ULN, ALT >2 × ULN, or AST >2 × ULN.
12. Hematocrit <20%, hemoglobin <70 g/L (<7 g/dL), or white blood count >15,000/μL.
13. Creatinine >1.5 × ULN.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10-09 (Estimated)

PRIMARY OUTCOMES:
The Number of participants with Drug-related SAE, All-cause SAE, Drug-related AESI, All-cause AESI. | up to 26 weeks
  To evaluate the safety of meplazumab in an adult population with uncomplicated, symptomatic P. falciparum infection
The Number of Participants discontinuation/ withdrawals due to AE | up to 26 weeks
  To evaluate the safety of meplazumab in an adult population with uncomplicated, symptomatic P. falciparum infection

CONTACTS AND LOCATIONS:
Locations (1):
- Kisumu County Referral Hospital, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No